CLINICAL TRIAL: NCT02465814
Title: A Randomized, Parallel-group, Double-blind Placebo-controlled and Open Label Active Controlled, Multi-center Study to Assess the Efficacy and Safety of Vilaprisan in Patients With Uterine Fibroids
Brief Title: Assess Safety and Efficacy of Vilaprisan in Patients With Uterine Fibroids
Acronym: ASTEROID 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17541; 2014-004221-41 (EudraCT Number)
Record Dates: First submitted 2015-05-22; First posted 2015-06-09 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Leiomyoma
Keywords: Uterine fibroids; Heavy Menstrual Bleeding
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — vilaprisan; ulipristal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm 1 - BAY1002670 + BAY1002670 (Experimental): Vilaprisan (BAY1002670) 2 mg once daily (12 weeks), Vilaprisan 2 mg once daily (12 weeks)
  Interventions: Drug: Vilaprisan (BAY1002670)
- Arm 2 - Placebo + BAY1002670 (Experimental): Placebo once daily (12 weeks), Vilaprisan 2 mg once daily (12 weeks)
  Interventions: Drug: Vilaprisan (BAY1002670
- Arm 3 - BAY1002670 + BAY1002670 (Experimental): Vilaprisan 2 mg once daily (12 weeks), treatment break, Vilaprisan 2 mg once daily (12 weeks)
  Interventions: Drug: Vilaprisan (BAY1002670
- Arm 4 - Placebo+BAY1002670 (Experimental): Placebo once daily (12 weeks), treatment break, Vilaprisan 2 mg once daily(12 weeks)
  Interventions: Drug: Vilaprisan (BAY1002670)
- Arm 5 - Ulipristal + Ulipristal (Active Comparator): Ulipristal 5 mg once daily (12 weeks), treatment break, Ulipristal 5 mg once daily (12 weeks)
  Interventions: Drug: Ulipristal
- Arm 6- Placebo + Ulipristal (Active Comparator): Placebo once daily (12 weeks), treatment break, Ulipristal 5 mg once daily (12 weeks)
  Interventions: Drug: Ulipristal
- Arm 7- Ulipristal + Placebo (Active Comparator): Ulipristal 5 mg once daily (12 weeks), treatment break, Placebo once daily (12 weeks)
  Interventions: Drug: Ulipristal

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — Vilaprisan 2 mg (12 weeks), Vilaprisan 2 mg (12 weeks)
  Arms: Arm 1 - BAY1002670 + BAY1002670
Drug: Vilaprisan (BAY1002670 — Placebo (12 weeks),Vilaprisan (12 weeks)
  Arms: Arm 2 - Placebo + BAY1002670
Drug: Vilaprisan (BAY1002670 — Vilaprisan 2 mg (12 weeks), treatment break, Vilaprisan 2 mg (12 weeks)
  Arms: Arm 3 - BAY1002670 + BAY1002670
Drug: Vilaprisan (BAY1002670) — Placebo (12 weeks), treatment break, Vilaprisan 2 mg (12 weeks)
  Arms: Arm 4 - Placebo+BAY1002670
Drug: Ulipristal — Ulipristal 5 mg (12 weeks), treatment break, Ulipristal 5 mg (12 weeks)
  Arms: Arm 5 - Ulipristal + Ulipristal
Drug: Ulipristal — Placebo (12 weeks), treatment break, Ulipristal 5 mg (12 weeks)
  Arms: Arm 6- Placebo + Ulipristal
Drug: Ulipristal — Ulipristal (12 weeks), treatment break, Placebo (12 weeks)
  Arms: Arm 7- Ulipristal + Placebo

SUMMARY:
The study is performed to assess the efficacy of Vilaprisan (BAY1002670) in patients with uterine fibroids compared to placebo and ulipristal. It is also aimed to evaluate the safety of vilaprisan in subjects with uterine fibroids. Further, data on population pharmacokinetic (PK)/ pharmacodynamic (PD) relationship for vilaprisan in subjects with uterine fibroids will be supplemented.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 to 50 years of age at the time of screening
* Diagnosis of uterine fibroid(s) documented by transvaginal or abdominal ultrasound at screening with at least 1 fibroid with largest diameter >/=3.0 cm
* Heavy menstrual bleeding (HMB) >80 mL documented by menstrual pictogram (MP) in a bleeding episode during the screening period. Women who did not suffer from perceived HMB during the 3 months prior to Visit 1 due to any effective medical treatment, e.g. with a hormonal contraceptive, are not considered appropriate candidates and should not undergo further screening procedures. Women suffering from perceived HMB despite medical treatment, e.g. with a hormonal contraceptive, are appropriate candidates for further screening, if rules on stopping prior medication are followed. Heavy menstrual bleeding /HMB) > 80 mL should be documented within 10 consecutive days.
* Good general health (except for findings related to uterine fibroids) as proven by medical history, physical and gynecological examinations, and laboratory test results
* Normal or clinically insignificant cervical smear not requiring further follow-up. Human papilloma virus (HPV) testing in subjects with atypical squamous cells of undetermined significance (ASCUS) can be used as an adjunctive test. Subjects with ASCUS can be included if they are negative for high-risk HPV strains.
* An endometrial biopsy performed during the screening period, without significant histological disorder such as endometrial hyperplasia (including simple hyperplasia) or other significant endometrial pathology.
* Use of an acceptable nonhormonal method of contraception (i.e. either male condom, cap, diaphragm or sponge, each in combination with spermicide) starting at the bleeding episode following the screening visit 1 (Visit 1) until the end of the study. This is not required if safe contraception is achieved by a permanent method, such as bilateral fallopian tube blockage of the subject or vasectomy of the partner(s).

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Uterine fibroid with largest diameter >10.0 cm
* Hypersensitivity to any ingredient of the study drugs
* Hemoglobin values </= 6 g/dL or any condition requiring immediate blood transfusion (subjects with hemoglobin values </=10.9 g/dL will be offered iron supplementation).
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Abuse of alcohol, drugs, or medicines (e.g. laxatives)
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results
* Undiagnosed abnormal genital bleeding.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Amenorrhea (yes/no) | From day 7 to day 84 of treatment.
  Defined as no scheduled or unscheduled bleeding/spotting after end of the initial bleeding episode until the end of the respective treatment period.

SECONDARY OUTCOMES:
Number of bleeding days | Up to 32 weeks
Time to onset of controlled bleeding | Up to 28 weeks
Percent change in volume of largest fibroid from baseline to end of treatment. | Baseline and up to 28 weeks
Endometrial histology | Baseline and up to 40 weeks
  (Frequency of the following categories: benign endometrium, endometrial hyperplasia, malignant neoplasm)
Endometrial thickness measured by transvaginal ultrasound. | Baseline and up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (54):
- Austria (4):
  - Villach, Carinthia
  - Graz, Styria
  - Innsbruck, Tyrol
  - Vienna, Vienna
- Belgium (3):
  - Tienen, Vlaams Brabant
  - Bruxelles - Brussel
  - Edegem
- Bulgaria (3):
  - Pleven
  - Sofia
  - Stara Zagora
- Czechia (6):
  - Brno
  - České Budějovice
  - Olomouc
  - Pilsen
  - Písek
  - Prague
- Finland (3):
  - Helsinki
  - Pori
  - Turku
- Germany (4):
  - Dresden, Saxony
  - Bernburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Hungary (3):
  - Budapest
  - Debrecen
  - Szentes
- Italy (3):
  - Modena, Emilia-Romagna
  - Cagliari, Sardinia
  - Catania, Sicily
- Vilnius, Lithuania
- Netherlands (4):
  - Almere Stad
  - Heerlen
  - Nieuwegein
  - Zwolle
- Norway (4):
  - Fredrikstad
  - Lørenskog
  - Nesttun
  - Stavanger
- Poland (4):
  - Bialystok
  - Lodz
  - Lublin
  - Warsaw
- Portugal (3):
  - Coimbra, Coimbra District
  - Lisbon, Lisbon District
  - Porto, Porto District
- Spain (3):
  - Barcelona, Barcelona
  - Aravaca, Madrid
  - Valencia, Valencia
- Sweden (2):
  - Stockholm
  - Umeå
- United Kingdom (4):
  - Harrow, London
  - London
  - Nottingham
  - Portsmouth

REFERENCES:
- [Derived] Gemzell-Danielsson K, Heikinheimo O, Zatik J, Poka R, Rechberger T, Hudecek R, Petersdorf K, Ramirez F, Faustmann T, Groettrup-Wolfers E, Seitz C. Efficacy and safety of vilaprisan in women with uterine fibroids: Data from the phase 2b randomized controlled trial ASTEROID 2. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:7-14. doi: 10.1016/j.ejogrb.2020.05.043. Epub 2020 May 31. PMID 32559602